CLINICAL TRIAL: NCT06715163
Title: Evaluation of the Safety and Tolerability of Three Doses of Diamine Oxidase (DAO) in Healthy Volunteers
Acronym: DAO-MAX2024
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotek (Industry)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DAO-MAX2024
Record Dates: First submitted 2024-11-19; First posted 2024-12-04 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Safety and Tolerability in Healthy Volunteers
Keywords: safety; tolerability; diamino oxidase; DAO; supplementation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose 1 (42mg) of DAO (Experimental): Lowest dose of DAO administered in this study
  Interventions: Dietary Supplement: Dose 1 (42mg) of DAO
- Placebo tablets (Placebo Comparator): placebo tablets
  Interventions: Dietary Supplement: Placebo
- Dose 2 (84mg) of DAO (Experimental): Medium dose of DAO administered in this study
  Interventions: Dietary Supplement: Dose 2 (84mg) of DAO
- Dose 3 (210mg) of DAO (Experimental): Highest dose of DAO administered in this study
  Interventions: Dietary Supplement: Dose 3 (210mg) of DAO

INTERVENTIONS:
Dietary Supplement: Dose 1 (42mg) of DAO — DAO extract is obtained from pea sprout dehydrated powder. Lowest dose of DAO administered in this study
  Other Names: diamino oxidase (DAO)
  Arms: Dose 1 (42mg) of DAO
Dietary Supplement: Placebo — Contains the same excipients as the DAO tablets but without the diamino oxidase content
  Arms: Placebo tablets
Dietary Supplement: Dose 2 (84mg) of DAO — DAO extract is obtained from pea sprout dehydrated powder. Medium dose of DAO administered in this study
  Arms: Dose 2 (84mg) of DAO
Dietary Supplement: Dose 3 (210mg) of DAO — DAO extract is obtained from pea sprout dehydrated powder. Highest dose of DAO administered in this study
  Arms: Dose 3 (210mg) of DAO

SUMMARY:
The main aim of this study is to evaluate the safety and tolerability of the product administered, of 3 different doses. Safety will be evaluated by recording and assessing adverse events, vital signs, laboratory tests and ECG. These assessments will be conducted during the study and at the end the study, following the study schedule and evaluation times. Since it is not absorbed and considering the conducted studies, 24 h are sufficient to analyse the safety and tolerability of the product. Safety will be assessed until the follow up visit, 6-8 days after product intake, to check possible adverse effects during that time.

ELIGIBILITY:
Inclusion Criteria:

1. - Subjects of either gender (male or female) aged ≥18 and ≤50 years at the time of the enrolment.
2. - Subjects free from organic or psychic conditions.
3. - No clinically significant abnormalities in medical records and physical examination at screening.
4. - No clinically significant abnormalities in haematology, biochemistry, serology (HBsAg, HCV antibodies, HIV antibodies) and urine drug results.
5. - Vital signs (blood pressure, respiratory rate, body temperature and pulse rate) and electrocardiogram record without clinically significant abnormalities.
6. - Body weight within the range (BMI ≥ 18.5 and ≤30.0 kg/m2) expressed as weight (kg) / height (m2).
7. - Free acceptance to participate in the study by obtaining signed informed consent form approved by the Ethics Committee of the Hospital (CEIm).

Exclusion Criteria:

1. - Background of allergy, idiosyncrasy or hypersensitivity to Investigational or any products or food
2. - Heavy consumers of stimulating drinks (>5 cups of coffee, tea, chocolate or cola drinks per day).
3. - Background History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 gr/day for men or 24 gr/day for women.
4. - Intake of any medication within 14 days prior to taking the study treatment (except for use of paracetamol short-term symptomatic treatments, according to the investigator criteria), or intake of over-the-counter products (including natural food supplements, vitamins and medicinal plants products) within 7 days prior taking the study treatment.
5. - Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results.
6. - Positive results for abuse drugs in urine test or ethanol in breath test (Day-1).
7. - Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, haematological, neurological disease or other chronic diseases.
8. - Females with positive results from the pregnancy test or breast-feeding.
9. - Smoking within 6 months prior to the study treatment phase (Period 1, Day -1). Smokers must refrain from any tobacco usage, including smokeless tobacco, nicotine patches, electronic cigarettes, etc. at least for 6 months prior to study treatment.
10. - Mentally or legally incapacitated at screening.
11. - Unwillingness or inability to follow the procedures outlined in the protocol.
12. - Volunteers who have difficulties in understanding the language in which the volunteer information is given.
13. - Any condition that, in the opinion of the investigator, may jeopardise the patient's well-being or the trial conduct according to the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Vital signs - blood pressure | from baseline (pre-dose) to 24 hours after treatment administration
  Systolic blood pressure (mmHg) and Diastolic blood pressure (mmHg)
Vital signs - Heart Rate | from baseline (pre-dose) to 24 hours after treatment administration
  Heart rate as bpm (beats per minute)
Vital signs - Respiratory Rate | from baseline (pre-dose) to 24 hours after treatment administration
  Respiratory rate as bpm
Vital signs - temperature | from baseline (pre-dose) to 24 hours after treatment administration
  Body temperature as ºC (Celsius degrees)
ECG - Ventricular Rate (HR) | from baseline (pre-dose) to 24 hours after treatment administration
  Electrocardiogram: Ventricular rate (bpm)
ECG - PR interval | from baseline (pre-dose) to 24 hours after treatment administration
  Electrocardiogram: PR interval (ms)
ECG - QRS interval | from baseline (pre-dose) to 24 hours after treatment administration
  Electrocardiogram: QRS interval (ms)
ECG - QT interval | from baseline (pre-dose) to 24 hours after treatment administration
  Electrocardiogram: QT interval (ms)
ECG - QTc interval | from baseline (pre-dose) to 24 hours after treatment administration
  Electrocardiogram: QTc interval through Bazett's formula (ms)
Laboratory analyses - Concentrations of Glucose, Urea, Triglycerides, Cholesterol measured as mmol/L | from baseline (pre-dose) to 24 hours after treatment administration
  BIOCHEMISTRY: Concentrations of Glucose, Urea, Triglycerides, Cholesterol measured as mmol/L
Laboratory analyses - Concentrations of Creatinine, Total Bilirubin measured as micromol/L | from baseline (pre-dose) to 24 hours after treatment administration
  BIOCHEMISTRY: Concentrations of Creatinine, Total Bilirubin measured as micromol/L
Laboratory analyses - Concentrations of GOT (AST), GPT (ALT), GGT, Alkaline Phosphatase measured as U/L | from baseline (pre-dose) to 24 hours after treatment administration
  BIOCHEMISTRY: Concentrations of GOT (AST), GPT (ALT), GGT, Alkaline Phosphatase measured as U/L.
Laboratory analyses - Concentrations of Albumin, Haemoglobin, CCMH measured as g/L. | from baseline (pre-dose) to 24 hours after treatment administration
  BIOCHEMISTRY: Concentrations of Albumin measured as g/L. HAEMATOLOGY: Concentrations of Haemoglobin, CCMH measured as g/L.
Laboratory analyses - Concentration of Haematocrit as L/L | from baseline (pre-dose) to 24 hours after treatment administration
  HAEMATOLOGY: Concentration of Haematocrit as L/L
Laboratory analyses - Concentration of Platelet count, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes measured as x10E9/L | from baseline (pre-dose) to 24 hours after treatment administration
  HAEMATOLOGY: Concentration of Platelet count, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes measured as x10E9/L.
Laboratory analyses | from baseline (pre-dose) to 24 hours after treatment administration
  SEROLOGY: HIV, HBV and HCV measured through ELISA analysis as presence or absence (positive or negative result).
Laboratory analyses | from baseline (pre-dose) to 24 hours after treatment administration
  SCREENING of DRUGS of ABUSE in URINE: ethanol, cannabis, amphetamines, cocaine, opiates and benzodiazepines measured as presence or absence (positive or negative result).
Incidence of adverse events | from baseline (pre-dose) to 24 hours after treatment administration
  Assessment through the opinion of the Investigator, who should consider if it is contraindicative to continue the volunteer's participation in the study if the volunteer experienced adverse events severe enough.

CONTACTS AND LOCATIONS:
Overall Officials: Pol Molina, PharmaD, Principal Investigator — Institut de Recerca Sant Pau
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Safety and tolerability of the treatments will be evaluated by assessing vital signs, laboratory analyses, ECG and incidence of AE.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: According to legislation